CLINICAL TRIAL: NCT02166632
Title: Prospective, Randomized Comparison of Postoperative Pain Control Results of Peri-articular Local Injection and Intra-capsular Injectinon of Bupivacaine Liposome Injectable Suspension After Total Knee Arthroplasty
Brief Title: Postoperative Pain Control Results Using Periarticular Versus Intra-capsular Injection of Bupivacaine Liposome Injectable Suspension in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Broward Health (Other)
Responsible Party: Principal Investigator, W Vincent Burke, MD, Orthopedic Surgeon, Broward Health, Broward Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BH130401
Record Dates: First submitted 2014-06-13; First posted 2014-06-18 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee arthroplasty; Exparel; Bupivacaine liposome; Total knee replacement; Pain control
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracapsular Injection (Experimental): Patients in the experimental group will undergo direct injection of ExparelTM into the knee joint; once the total knee replacement (arthroplasty) has been completed, patients will receive a given amount of ExparelTM administered during surgery into the joint where the knee replacement (arthroplasty) (TKA) was performed.
  Interventions: Procedure: Intracapsular Injection
- Periarticular Injection (Active Comparator): Patients in this group will undergo local injection of ExparelTM to help to reduce post-surgery pain. Once the total knee replacement (arthroplasty) has been completed, patients in this group will receive a given amount of ExparelTM administered during surgery into the soft tissues around the bone where the knee replacement (arthroplasty) (TKA) was performed.
  Interventions: Procedure: Periarticular Injection

INTERVENTIONS:
Procedure: Intracapsular Injection — The amount of bupivacaine liposome (ExparelTM) will be injected directly into the joint capsule (intracapsular injection), effectively "bathing" the joint in the medication.
  Other Names: Intracapsular injection of bupivacaine liposome (ExparelTM)
  Arms: Intracapsular Injection
Procedure: Periarticular Injection — The amount of bupivacaine liposome (ExparelTM) will be injected periarticulary, via 9 standard periarticular tissue sites around the joint
  Other Names: Periarticular injection of bupivacaine liposome (ExparelTM)
  Arms: Periarticular Injection

SUMMARY:
The purpose of this study is to determine quantitative and qualitative differences in post-operative pain relief for patients undergoing primary total knee arthroplasty (TKA) who receive administration of a newly approved, long acting local anesthetic branded as ExparelTM (bupivacaine liposome injectable suspension) introduced by one of two different administration methods.

Group 1 would receive a predetermined and standardized dose of ExparelTM introduced directly into the joint capsule at the conclusion of the surgery, effectively bathing the joint in anesthetic solution.

Group 2 would receive the same predetermined and standardized dose of ExparelTM as a local infiltration anesthetic (LIA) by injecting it into the periarticular tissues in nine (9) standard sites at the conclusion of the surgery.

DETAILED DESCRIPTION:
This study is being done to determine if a difference exists between two methods of intraoperative (during surgery) administration of a long-acting local anesthetic (pain relief).

Local pain relief medications are accepted as standard of care as a part of a comprehensive plan for pain relief following a total knee replacement (arthroplasty) (TKA). We expect that the addition of ExparelTM to the usual post-surgery pain control medicines and procedures will result in less need for additional pain medication. It is possible that local injection into the tissue around the total knee replacement joint (periarticular tissues) may provide more effective pain relief than injection directly into the joint (intracapsular) itself, or vice versa. It is also possible that pain relief with either method is approximately equivalent. On the day of surgery, each patient will undergo total knee arthroplasty and cared for utilizing the standard protocol for all patients that undergo total knee arthroplasty at Broward Health Medical Center.

Patients in Group 1 will receive the same amount of ExparelTM injected intracapsularly. Those in is Group 2 will receive a standardized medication regimen including ExparelTM by local infiltration into the periarticular tissues at the conclusion of their TKA procedure. Study participants will undergo injection in this manner until the conclusion of the study.

All subjects will be provided the same methods of postoperative pain control following their TKA surgery as those patients not enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over the age of 18
* Patients must have a preoperative diagnosis of osteoarthritis of the knee requiring total knee arthroplasty

Exclusion Criteria:

* Allergy to ExparelTM or certain other local anesthetic agents
* Pregnant females or females who think they may become pregnant
* Markedly abnormal kidney function or renal disease
* History of substance abuse
* History of chronic pain requiring medication
* Had a previous total knee arthroplasty on the same knee which is being replaced (revision total knee arthroplasty)
* Had a previous partial knee arthroplasty, such as a unicompartmental knee arthroplasty on the same knee (also a revision total knee arthroplasty)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale for Pain | 8 weeks pre-surgery (Baseline/Day 0) and every day for 1 week, post-surgery (Day 1, 2, 3, 4, 5, 6, 7)
  Pre-Surgical visual analog scale for pain will be administered up to 2 months pre-surgery.
  Post-Surgical visual analog scales will be administered as a "pain journal" in which patients will record their level of pain twice a day, once in the morning, and once in the evening for 1 week.

SECONDARY OUTCOMES:
Change in Oxford Knee Score | 8 weeks pre-surgery (baseline) and 4 weeks post surgery (Day 28)
  Pre-surgical oxford knee questionnaires will be administered up to 2 months pre-surgery. Post-surgical questionnaires will be administered at the patient's first follow-up office visit, approximately 4 weeks post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: William V Burke, M.D., Principal Investigator — Broward Health
Locations (1):
- Broward Health Sports Medicine, Fort Lauderdale, Florida, United States